CLINICAL TRIAL: NCT03940911
Title: Fatigue and Skeletal Muscle Impact in Severe Axial Spondyloarthritis
Acronym: Famuspa
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 7439
Record Dates: First submitted 2019-05-06; First posted 2019-05-07 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Spondyloarthritis, Axial; Fatigue; Exercise Capacity
Keywords: Axial spondylarthritis; Fatigue; Targeted therapy; Exercise capacity; Sarcopenia
MeSH Terms: conditions — Axial Spondyloarthritis; Fatigue; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Targeted therapy and severe fatigue (FSS) (Other): See bellow (section "Interventions") the full description for
  * Measurement of aerobic exercise on cycloergometer
  * Measurement of muscle mass by two-photon absorptiometry: specific study
  * Measurement of Isometric Muscle Strength
  * Blood sampling for measurement of cytokine levels in the blood
  * Measurement of sedentarity
  * Psychological impact
  * Fatigue measurement
  Interventions: Other: Measurement of aerobic exercise on cycloergometer
- Targeted therapy and mild fatigue (FSS <4) (Other): See bellow (section "Interventions") the full description for
  * Measurement of aerobic exercise on cycloergometer
  * Measurement of muscle mass by two-photon absorptiometry: specific study
  * Measurement of Isometric Muscle Strength
  * Blood sampling for measurement of cytokine levels in the blood
  * Measurement of sedentarity
  * Psychological impact
  * Fatigue measurement
  Interventions: Other: Measurement of aerobic exercise on cycloergometer

INTERVENTIONS:
Other: Measurement of aerobic exercise on cycloergometer — The incremental effects tests will be performed in a service specialized in the exploration of the exercise (physiology or cardiology according to the centers) in a spacious and air-conditioned room, in the presence of a medical specialist. exercise and close to the resuscitation equipment.
  Before the test, weight and height will be collected. Information on the conduct of the test will be given to the patient. A multi-derivation ECG recording will be detected throughout the duration of the test and followed by a physician experienced in the ECG effort.
  O2 saturation by oximetry of hens will be recorded continuously. Blood pressure will be recorded at each level. The collection of expired gases in the face mask whose tightness will be verified to measure the fractions inspired and expired in O2 and CO2 (Sensor Medics Vmax229, Yorba Linda, CA, USA) and calculations VO2 max and VCO2.
  Maximal power (W max) will be recorded. Patients will be encouraged during the test.

SUMMARY:
Axial spondyloarthropathy (SpA) is the most common inflammatory rheumatism (1% of the general population) with important medico-economic consequences.

Fatigue is a major feature of SA. It can be defined as a feeling of reduced muscle capacity, lack of energy and exhaustion. The fatigue reaches an abnormally high level (fatigue severity score (FSS) ≥4, called severe fatigue in this protocol) in more than two thirds of patients with SA.

Skeletal muscle repercussions are present during SA. It is characterized by a decrease in exercise capacity independently of pain and ankylosis but is associated with a decrease in strength and muscle mass, the importance of which varies from one study to another.

The link between fatigue (subjective sensation) and the skeletal muscular impact (objective) of SA has never been studied.

DETAILED DESCRIPTION:
This work will:

1. Study for the first time the implication of the objective skeletal muscular impact in fatigue during SA.
2. Better characterize the skeletal muscle impact of SA;
3. Characterize the evolution of the fatigue and the muscular impact under targeted therapy

ELIGIBILITY:
Inclusion criteria:

* Axial SA according to the ASAS criteria;
* Targeted therapy naïve patients
* Indication to start a targeted therapy;
* Initiation of targeted therapy ≤ 15 days before inclusion
* ≥ 18 years old, no upper age limit;
* Subject affiliated to a social health insurance reimbursement;
* Subject able to understand the aims and risks of the research and having signed a dated and informed consent
* Subject informed of the results of the preliminary medical examination
* Woman in childbearing age: negative beta-HCG test and effective contraception;
* Sufficient understanding of French to follow the protocol.

Exclusion criteria:

* Targeted therapy in progress for > 15 days prior to inclusion
* Contraindication to the use of targeted therapy
* Systemic corticosteroids in the 15 days preceding the V0 visit
* Associated extramuscular inflammatory disease (s) (excluding ocular and cutaneous involvement) eg chronic inflammatory bowel disease
* Associated fibromyalgia (Questionnaire score FiRST ≥5) achieved during the V0 visit
* History of coronary artery disease: exercise angina, acute coronary syndrome and / or coronary angioplasty,
* History of lower extremity arterial disease: vascular claudication and / or lower extremity angioplasty
* COPD
* Neuromuscular pathology
* Insufficiency of organ (renal, hepatic pulmonary heart)
* Sleep apnea
* Impossibility of giving the subject informed information (subject in emergency situation, difficulties in understanding the subject, etc.)
* Subject under the protection of justice
* Subject under guardianship or curatorship
* Breastfeeding
* Pregnancy
* Subject in exclusion period defined by another clinical study or participating in a study likely to impact the results of the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Oxygen consumption capacity | At inclusion
  Maximum oxygen consumption capacity on cycloergometer during an incremental effort until exhaustion (VO2 max)

IPD SHARING:
Plan to Share IPD: No